CLINICAL TRIAL: NCT00130377
Title: Biological Cell Therapy for the Treatment of Patients With Thoracic & Cardiovascular Disease
Brief Title: Evaluation of the Treatment of Thoracic & Cardiovascular Disease With Biological Therapy: ClinicalCellRegistry.Com
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amit N. Patel MD MS (Other)
Responsible Party: Sponsor-Investigator, Amit N. Patel MD MS, Amit Patel, Amit, Patel N, M.D.
Organization: Amit, Patel N, M.D. (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0506137
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Cardiovascular System Diseases (& [Cardiac])
Keywords: Stem Cell; Heart; Lung; Vascular; cell therapy registry
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cell therapy (Experimental): Patient receiving active biologic
  Interventions: Biological: cell therapy
- control (Placebo Comparator): Patient receiving placebo or standard of care
  Interventions: Biological: cell therapy

INTERVENTIONS:
Biological: cell therapy — autologous or allogeneic cells

SUMMARY:
This is the clinical registry of cell based therapies that is available to researchers around the world. The registry is web based. All researches must provide IRB approval to the coordinating site- University of Utah in order to obtain access to the registry. The are predetermined case report forms for cardiovascular diseases that are currently in clinical trials- including demographics, safety, and possible efficacy end-points. All investigators have access to their own data. The servers are U.S. HIPPA compliant and protected with secure back-up.

DETAILED DESCRIPTION:
The clinical cell registry includes data on thoracic and cardiovascular diseases including:

Acute myocardial infarction, Chronic Angina, Heart Failure, Wound Healing including Sternal, Peripheral Arterial Disease, Critical Limb Ischemia, Type 2 Diabetes, COPD, Asthma. Neurological disorders registry is available to specifics sites if requested. Our own biological data at the University of Utah including co-localized data with Society of Thoracic Surgeons also is a part of this program. Cell based therapies that are autologous and allogeneic are included in the registry

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old
* Approved consent to be enrolled in trial/registry

Exclusion Criteria:

* Prior malignancy in the 5 years before treatment in this study (other than curatively treated carcinoma in-situ of the cervix or non-melanoma skin cancer)
* Inability or unwillingness to comply with the treatment protocol, follow-up, research tests, or give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2002-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Safety - MACE - Death, Readmission, Reintervention | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amit N. Patel, MD, MS, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Lin F, Josephs SF, Alexandrescu DT, Ramos F, Bogin V, Gammill V, Dasanu CA, De Necochea-Campion R, Patel AN, Carrier E, Koos DR. Lasers, stem cells, and COPD. J Transl Med. 2010 Feb 16;8:16. doi: 10.1186/1479-5876-8-16. PMID 20158898
- [Background] Bruckner BA, Ghodsizad A, Loebe M, Beyer E, Ramchandani M, Ruhparwar A, Karck M, Burchardt ER, Patel AN, Reardon M. Surgical stem cell therapy for advanced heart failure patients. Methodist Debakey Cardiovasc J. 2009;5(2):13-7. doi: 10.14797/mdcj-5-2-13. No abstract available. PMID 20073160
- [Background] Patel AN, Sherman W. Cardiac stem cell therapy: advances from 2008. Cell Transplant. 2009;18(3):243-4. doi: 10.3727/096368909788534960. No abstract available. PMID 19558772
- [Background] Sherman W, Mazouz C, Deans R, Patel AN. Commercialization of trials for peripheral artery disease. Cytotherapy. 2011 Nov;13(10):1157-61. doi: 10.3109/14653249.2011.620795. No abstract available. PMID 21999371
- [Background] Benoit E, O'Donnell TF Jr, Iafrati MD, Asher E, Bandyk DF, Hallett JW, Lumsden AB, Pearl GJ, Roddy SP, Vijayaraghavan K, Patel AN. The role of amputation as an outcome measure in cellular therapy for critical limb ischemia: implications for clinical trial design. J Transl Med. 2011 Sep 27;9:165. doi: 10.1186/1479-5876-9-165. PMID 21951607
- [Background] Tuma J, Fernandez-Vina R, Carrasco A, Castillo J, Cruz C, Carrillo A, Ercilla J, Yarleque C, Cunza J, Henry TD, Patel AN. Safety and feasibility of percutaneous retrograde coronary sinus delivery of autologous bone marrow mononuclear cell transplantation in patients with chronic refractory angina. J Transl Med. 2011 Oct 26;9:183. doi: 10.1186/1479-5876-9-183. PMID 22029669
- [Result] Patel AN, Geffner L, Vina RF, Saslavsky J, Urschel HC Jr, Kormos R, Benetti F. Surgical treatment for congestive heart failure with autologous adult stem cell transplantation: a prospective randomized study. J Thorac Cardiovasc Surg. 2005 Dec;130(6):1631-8. doi: 10.1016/j.jtcvs.2005.07.056. Epub 2005 Oct 26. PMID 16308009
- [Result] Patel AN, Mittal S, Turan G, Winters AA, Henry TD, Ince H, Trehan N. REVIVE Trial: Retrograde Delivery of Autologous Bone Marrow in Patients With Heart Failure. Stem Cells Transl Med. 2015 Sep;4(9):1021-7. doi: 10.5966/sctm.2015-0070. Epub 2015 Jul 27. PMID 26217065
- [Result] Patel AN, Silva F, Winters AA. Stem cell therapy for heart failure. Heart Fail Clin. 2015 Apr;11(2):275-86. doi: 10.1016/j.hfc.2014.12.006. PMID 25834975
- [Derived] Patel AN, Selzman CH, Kumpati GS, McKellar SH, Bull DA. Evaluation of autologous platelet rich plasma for cardiac surgery: outcome analysis of 2000 patients. J Cardiothorac Surg. 2016 Apr 12;11(1):62. doi: 10.1186/s13019-016-0452-9. PMID 27068030